# Statistical Analysis Plan for Protocol

207196

A Randomized, Parallel-group, Evaluator-blind, No-treatment and Positive-controlled, Single-site, Proof-of-concept Clinical Study to Evaluate the Cosmetic Benefit Provided by 8 Weeks of Twice-daily Topical Application of a Developmental Moisturizing Cream with Niacinamide in Healthy Subjects with Sensitive, Oily, Blemish-prone Skin

## NCT03093181

#### GlaxoSmithKline Consumer Healthcare

980 Great West Road, Brentford, Middlesex, TW8 9GS, UK.

1. Statistical Analysis Plan approval date: 19-SEP-2017
2. Final Amendment to Statistical Analysis Plan approval date: 20-DEC-2017

Copyright: GlaxoSmithKline. This document contains confidentiality statements that are not relevant for this publicly available version



#### STATISTICAL REPORTING AND ANALYSIS PLAN

A randomised, parallel-group, evaluator-blind, no-treatment and positive controlled, single-site, proof of concept clinical study to evaluate the cosmetic benefit provided by 8 weeks of twice-daily topical application of a developmental moisturising cream with niacinamide in healthy subjects with sensitive, oily, blemish-prone skin

Protocol Number: 207196

Phase: NA

This document contains confidentiality statements that are not relevant for this publicly available version.

Property of GSK Consumer Healthcare
Confidential

May not be used, divulged, published or otherwise disclosed without the consent of GSK

Template Version Effective: 15-Jul-2017

Page 1 of 62

## **Document History**

| Document | Version Date | Summary of Changes (New analysis or Change in planned analysis) |
|---|---|---|
| Original Analysis Plan | 19-Sept-2017 | Not applicable (N/A) |

| 18 | | conter | <b>11S</b><br>tory | 2 |
|---|---|---|---|---|
| | | | nts | |
| | | | шо | |
| 1 | | • | ey Protocol Information | |
| 1 | 1.1 | - | Design | |
| | 1.2 | • | Objectives | |
| | 1.3 | • | ents | |
| | 1.4 | | Size Calculation | |
| 2 | | - | sessize Caretaidon | |
| _ | 2.1 | • | Analysis | |
| | 2.2 | | nalyses | |
| 3 | | | for data analyses and Data Handling Conventions | |
| 5 | 3.1 | | e Definition | |
| | 3.2 | | ups/Stratifications | |
| | 3.3 | _ | bints and Visit Windows | |
| 4 | | • | omts and visit windows | |
| • | 4.1 | • | tions for Analysis | |
| | 7.1 | 4.1.1 | Subject Disposition | |
| | | 4.1.2 | Protocol Deviations | |
| | | 4.1.3 | Analysis Populations | |
| | 4.2 | | Demographics and Other Baseline Characteristics | |
| | 7.2 | 4.2.1 | Demographic Characteristics | |
| | | 4.2.2 | General Medical History | |
| | 4.3 | | ents (Study Product, Rescue Medication, other Concomitant | 13 |
| | 1.5 | | ies, Compliance) | 13 |
| | | 4.3.1 | Study Product Compliance and Exposure | 13 |
| | | 4.3.2 | Prior and Concomitant Medication | |
| | 4.4 | Analysi | is of Efficacy | 14 |
| | | 4.4.1 | Primary Efficacy Endpoint | 14 |
| | | 4.4.2 | Secondary Efficacy Variables | |
| | | 4.4.3 | Handling of Missing Values/Censoring/Discontinuations | |
| | 4.5 | Analysi | is of Secondary Objectives | |
| | | 4.5.1 | Efficacy | |
| | | | - · | |



| | | 4.5.2 | Pharmacokinetic (Secondary) | 17 |
|----|--------|------------|----------------------------------------------|----|
| | 4.6 | Analys | sis of Safety | 17 |
| | | 4.6.1 | Adverse Events and Serious Adverse Events | 17 |
| | | 4.6.2 | Other Safety Variables | 17 |
| | 4.7 | Analys | sis of Other Variables | 17 |
| 5 | Chan | ges to the | e Protocol Defined Statistical Analysis Plan | 17 |
| At | tachme | nt 1: List | of Data Displays | 19 |
| At | tachme | nt 2: Ten | nplate for Tables, Figures and Listings | 20 |

## Glossary

| AE | Adverse Event |
|--------|----------------------------------------------|
| ANCOVA | Analysis of covariance |
| BDRM | Blind Data Review Meeting |
| CI | Confidence Interval |
| ITT | Intent-to-Treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PP | Per Protocol |
| RAP | Statistical Reporting and Analysis Plan |
| RH | Relative Humidity |
| RLR | Review Listing Requirement |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Event |

The purpose of this Statistical Reporting and Analysis Plan is to describe the planned analyses and outputs to be included in the Clinical Study Report for Protocol 207196.

#### 1 Summary of Key Protocol Information

This randomised, parallel-group, evaluator-blind, no-treatment and positive controlled, single-site, proof of concept clinical study is designed to evaluate the cosmetic benefit provided by 8 weeks of twice-daily topical application of a developmental moisturising cream with niacinamide in healthy subjects with sensitive, oily, blemish-prone skin.

General safety and tolerability will be assessed based on the frequency and severity of Adverse Events (AEs).

#### 1.1 Study Design

This randomised, parallel-group, evaluator-blind, no-treatment and positive controlled, single-site, proof of concept clinical study follows the study schedule below.

| Procedure/Assessment | Visit 1<br>Day-7 to -5 | Visit 2<br>Day 1 | Visit 3<br>Day 8 ± 1 | Visit 4<br>Day 29 ± 2 | Visit 5<br>Day 57 ± 2 |
|---|---|---|---|---|---|
| | Screening<br>/Washout | Baseline | 1 Week of<br>Application | 4 Week of<br>Application | 8 Week of<br>Application |
| Inform Consent | ✓ | | | | |
| Demographics | ✓ | | | | |
| Medical History | ✓ | | | | |
| Current / Concomitant Medication | ✓ | ✓ | ✓ | ✓ | ✓ |
| Adverse Events | | ✓ | ✓ | ✓ | ✓ |
| Diary Review (Compliance) <sup>1</sup> | | ✓ | ✓ | ✓ | ✓ |
| Continued Eligibility | | ✓ | ✓ | ✓ | ✓ |
| Fitzpatrick Skin Type Assessment | ✓ | | | | |
| Evaluator Assessment of Blemish Counts <sup>2</sup> | ✓ | <b>√</b> <sub>4</sub> | ✓ | ✓ | ✓ |
| Forehead Sebumeter Measurement <sup>3</sup> | ✓ | <b>√</b> <sub>4</sub> | ✓ | ✓ | ✓ |
| Inclusion / Exclusion Criteria | ✓ | <b>√</b> <sub>5</sub> | | | |
| Subject Eligibility | ✓ | ✓ | | | |
| Washout Cleanser and Diary Dispensing | ✓ | | | | |
| Randomisation | | ✓ | | | |

| Corneometer Measurements <sup>3</sup> | <b>√</b> <sub>4</sub> | ✓ | ✓ | ✓ |
|---|---|---|---|---|
| Image Capture | $\checkmark_4$ | | | ✓ |
| Washout Cleanser return and Products Dispensing | ✓ | | | |
| Sebumeter Kinetic Measurements <sup>3,9</sup> | <b>✓</b> | ✓ | ✓ | ✓ |
| Supervised Product Application <sup>6</sup> | <b>✓</b> | ✓ | ✓ | |
| Acute Corneometer Measurements | <b>√</b> 7 | | | |
| Products and Diary Return | | | | ✓ |
| Subject Discharge from Study | | | | <b>✓</b> |
| Lay Person Assessment of Overall Appearance of Blemishes (Photographs) <sup>5</sup> | | | | ✓ |

- 1. Evaluators must be blinded to diary review.
- 2. Blind evaluator assessment of papules and pustules, to be counted separately for the face, chin and cheeks.
- 3. Time Subjects must also acclimatize for a minimum of 30 minutes in a temperature ( $20 \pm 1$  degrees Celsius ( $^{\circ}$ C)) and humidity ( $50 \pm 10\%$  Relative Humidity (RH)) controlled room prior to any instrumental measurement being taken.
- 4. Baseline measurements (prior to any product application).
- 5. Only the inclusion and exclusion criteria in Appendix 2 will be reviewed at this visit.
- 6. Subjects randomised to positive control regimen will apply the positive control cleanser and positive control cream. Subjects randomised to the test product regimen will apply the standard cleanser and test product. Subjects randomised to the no treatment regimen will apply the standard cleanser only. Test product application will be overseen by a member of the study team who must not be involved in any clinical or instrumental assessment which could influence the study outcome.
- 7. Acute Corneometer assessments will be taken 1 hour  $\pm$  15 MINUTES, 3 hours  $\pm$  15 MINUTES and 8 hours  $\pm$  15 MINUTES after application of the cream for subjects randomised to the test product and positive control regimens and after cleansing for subjects randomised to the untreated regimen.
- 8. Lay person assessment of overall appearance of blemishes (Photographs) will take place after the completion of the clinical study.
- 9. Sebumeter kinetic measurements will be taken  $5\pm1$  minutes and  $90\pm5$  minutes after forehead cleansing.

#### 1.2 Study Objectives

| Objectives | Endpoints |
|---|---|
| Primary | |
| Evaluation of skin moisturisation | Corneometer values at 8 hours on Day 1 |
| (change from baseline) compared to | |
| no treatment | |
| Secondary | |
| Evaluation of skin moisturisation | Corneometer values at 1 hour on Day 1, 3 hours |
| (change from baseline) compared to | on Day 1, 1 week, 4 weeks and 8 weeks |
| no treatment | |
| Evaluation of the overall appearance | Lay person assessment of the appearance |

| Objectives | Endpoints |
|---|---|
| of blemishes (change from baseline) | of blemishes by photographic assessment |
| compared to no treatment | at 8 weeks |
| | Evaluator assessment blemish count (sum of papules and pustules at forehead, chin and cheeks) at 1, 4 and 8 weeks |
| | Evaluator assessment of individual blemish count (individual count of papules and pustules at the forehead, chin and cheeks) at 1, 4 and 8 weeks |
| Evaluation of skin oiliness | Sebumeter values at 1, 4 and 8 weeks |
| improvement (change from baseline) | |
| compared to no treatment | Sebum excretion rate at 1, 4 and 8 weeks |
| To evaluate the safety of the test product | Frequency and severity of adverse events |

#### 1.3 Treatments

| | Washout/<br>Standard<br>Cleanser | Test Product | Positive<br>Control<br>Cleanser | Positive<br>Control<br>Moisturiser |
|---|---|---|---|---|
| Product<br>Name | Simple Kind to<br>Skin<br>Moisturising<br>Facial Wash | Moisturising<br>Cream with<br>Niacinamide | Neutrogena<br>Visibly Clear<br>Spot Clearing<br>Facial Wash | Vivatinell<br>Acnecinamide<br>Gel Cream |
| Product<br>Formulation<br>Code (MFC) | Commercially<br>Available (UK) | CCI | Commercially<br>Available (UK) | Commercially<br>Available<br>(Turkey) |
| Application<br>Quantity | Approx. 0.6 g | Approx. 0.6 g | Approx. 0.6 g | Approx. 0.6 g |
| Application<br>Instructions | Use twice daily<br>(morning and<br>night) with at<br>least 8 hours | Use twice<br>daily (morning<br>and night) with<br>at least 8 hours | Use twice daily<br>(morning and<br>night) with at<br>least 8 hours | Use twice daily<br>(morning and<br>night) with at<br>least 8 hours |
| | between product applications. | between<br>product | between product applications. | between product applications. |

| Washout/<br>Standard<br>Cleanser | Test Product | Positive<br>Control<br>Cleanser | Positive<br>Control<br>Moisturiser |
|---|---|---|---|
| Wet your face | applications. | Wet your face | Apply a |
| and hands with | Dispense two | and hands with | peasized |
| water. Dispense | pumps of | water. Dispense | quantity to your |
| the product into | product onto | the product into | whole face, |
| your hands and | your fingertips | your hands and | covering all |
| apply to the | and apply to | apply to the | blemishes. |
| face. Massage | your whole | face. Massage | Avoid contact |
| gently. Rinse | face, covering | gently. Rinse | with eyes. If |
| with water and | all blemishes. | with water and | contact occurs, |
| pat dry. Avoid | Avoid contact | pat dry. Avoid | rinse thoroughly |
| contact with | with eyes. If | contact with | with water. |
| eyes. If contact | contact occurs, | eyes. If contact | |
| occurs, rinse | rinse | occurs, rinse | |
| thoroughly with | thoroughly | thoroughly with | |
| water. | with water. | water. | |

### 1.4 Sample Size Calculation

Approximately 200 female subjects aged 18-45 with self-assessed sensitive skin and a minimum of 8 and a maximum of 25 facial blemishes (papules and pustules, excluding the nose) will be screened to randomise 132 healthy subjects, to ensure approximately 40 subjects in the test product regimen, 40 subjects in the no treatment regimen and 40 subjects in the positive control regimen complete the study (Assuming a 10% dropout rate). Randomisation will be stratified by age (<21 years old, ≥21 years of age).

The sample size was based on clinical considerations. In a previous study of a cosmetic product, counts of papules and pustules decreased from a baseline mean of 27.6 to a mean of 13.5 at Week 8 (ref. Shalita 1995 IJD). With 40 subjects in both the test product and notreatment regimens, a difference between groups at least 60% the magnitude of the standard deviation (assumed equal for both groups) would be detectable at two-sided alpha=0.05 with approximately 80% power.

#### 2 Planned Analyses

#### 2.1 Interim Analysis

No interim analysis is planned.

#### 2.2 Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and database has been locked.
- 3. All criteria for unblinding the randomisation codes have been met and the randomisation codes have been distributed.

# 3 Considerations for data analyses and Data Handling Conventions

#### 3.1 Baseline Definition

For all endpoints the baseline value will be the latest before test product or positive control product for subjects randomised to the test regimen and positive control regimen, and before baseline cleansing for subjects randomised to the untreated regimen.

#### 3.2 Subgroups/Stratifications

Eligible subjects will be stratified by age (<21 years, ≥21 years) when randomised into treatments. There are therefore two strata in this study:

- Stratum1: Subjects of age<21 years;
- Stratum2: Subjects of age ≥21 years.

#### 3.3 Timepoints and Visit Windows

Deviations from the scheduled assessment times should be avoided or kept to a minimum as possible. Any deviation will be noted in the blinded data review before database lock and subjects may be considered for exclusion from the per protocol population.

The following are the assessment time windows.

| Visit | Time window |
|---------|-------------------------------------------------------------------|
| Visit 2 | 5-7 days after Visit 1. Visit 2 is baseline and counted as Day 1. |
| Visit 3 | Day 8 ± 1 Day |

| Visit | Time window |
|---------|---------------------|
| Visit 4 | $Day 29 \pm 2 Days$ |
| Visit 5 | Day 57 ± 2 Days |

Acute corneometer assessments will be taken 1 hour  $\pm$  15 MINUTES, 3 hours  $\pm$  15 MINUTES and 8 hours  $\pm$  15 MINUTES after application of the cream for subjects randomised to the test product and positive control regimens and after cleansing for subjects randomised to the untreated regimen.

Sebumeter kinetic measurements will be taken  $5 \pm 1$  minutes and  $90 \pm 5$  minutes after forehead cleansing.

#### 4 Data Analysis

Data analysis will be performed by inVentiv Health Clinical. Prior to database closure a Blind Data Review Meeting (BDRM) will be conducted in which various aspects of the trial will be discussed and agreed. The statistical analysis software used will be SAS version 9.4.

Unless otherwise described below, all listings will be produced for all randomized subjects.

#### 4.1 Populations for Analysis

Tables described in this section will be produced for all randomised subjects, unless otherwise specified.

#### 4.1.1 Subject Disposition

Screen failures will be defined as subjects who consent to participate in the study but are never subsequently randomised. A summary will be provided of the number of subjects screened and the number of screen failures.

Subject disposition will be summarised as the number and percentage of subjects (out of the number of randomised subjects) who complete the study, with the number who discontinue broken down by reason for discontinuation (Table 14.1.1). The table will also summarise the number and percent of subjects assigned to each analysis population (defined in Section 2.1.3). The summary will be presented by treatment and overall.

Subject disposition will be listed for randomised subjects (Listing 16.2.1.1) and non-randomised subjects (Listing 16.2.1.2) separately.

#### 4.1.2 Protocol Deviations

Protocol deviations will be tracked by the study team throughout the conduct of the study. All deviations will be reviewed prior to unblinding and closure of the database to ensure all important violations are captured and categorised.

Major deviations identified as liable to influence the efficacy outcome will include follows:

- Deviation from the inclusion/exclusion criteria
- Use of prohibited medication
- Not receiving randomised treatment

Further deviations liable to influence the efficacy outcome will be given in the "Review Listing Requirement (RLR)" document and major deviations will be identified in blinded data review stage. The number and percentage of subjects with any major protocol deviations and with each type of major protocol deviations will be presented by treatment (Table 14.1.2) and listed (Listing 16.2.2.1). Any minor protocol deviations will be listed similarly (Listing 16.2.2.2).

#### 4.1.3 Analysis Populations

Six analysis populations are defined.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Screened | All subjects those who are screened | Disposition |
| Subjects | | |
| Randomised | All subjects who are randomised and may or | Protocol deviations |
| | may not receive the application of the study | |
| | products. | |
| Safety | Safety population includes all subjects who | Safety analysis |
| | are randomised and receive at least one dose | |
| | of study product. For the no-treatment | |
| | regimen, this will include any use of the | |
| | cleanser post-randomisation. | |
| Intent-to-Treat | The 'Intent to treat' (ITT) population | Efficacy analysis |
| (ITT) | includes all subjects who are in safety | |
| | population and have at least one post | |
| | baseline efficacy assessment. | |
| Per-Protocol | The Per Protocol (PP) population will consist | Efficacy analyses for |
| (PP) | of the subset of ITT subjects which excludes | corneometry and |
| | those subjects with major protocol | blemish count will also |
| | deviations. | be performed on the PP |
| | | population |

The numbers of subjects included in each of the analysis populations, and the number excluded from each population broken down by the reason for exclusion will be presented (Table 14.1.3). Subjects excluded from any of the analysis populations will be listed (Listing 16.2.3.1).

#### 4.2 Subject Demographics and Other Baseline Characteristics

#### 4.2.1 Demographic Characteristics

Categorical demographic variables include sex, race and Fitzpatrick type. These variables will be summarised by the number and percentage of subjects with each relevant characteristic (Table 14.1.4.1 for the Safety population, Table 14.1.4.2 for the ITT population and Table 14.1.4.3 for the PP population). Age will be summarised by the mean, standard deviation (SD), median, minimum and maximum values. Baseline stratification will also be summarised by the number and percentage of subjects in each stratum. All summaries will be presented by treatment, and overall. All demographic information will be listed (Listing 16.2.4.1).

#### 4.2.2 General Medical History

Medical history data will be listed in Listing 16.2.4.2 with start date and end date or ongoing at the start of study drug. A data listing will also be produced for evaluation of protocol violations at the blinded data review stage.

# 4.3 Treatments (Study Product, Rescue Medication, other Concomitant Therapies, Compliance)

#### 4.3.1 Study Product Compliance and Exposure

Study product compliance (using study products twice daily) will be listed (Listing 16.2.5.1) and checked at the blinded data review stage for evaluation of protocol violations. A compliance summary table will be provided for ITT population (Table 14.2.1).

#### 4.3.2 Prior and Concomitant Medication

Prior and concomitant medication/non-drug treatments data will be listed (Listing 16.2.5.2, 16.2.5.3). Prior medications are defined as those stopped before the baseline administration of the study products. Concomitant medications are defined as those ongoing or started on or after the baseline administration of the study products.

A data listing will also be produced for evaluation of protocol violations at the blinded data review stage.

#### 4.4 Analysis of Efficacy

Statistical testing of all endpoints in this study will be conducted at unadjusted two-sided significance level of 0.05. The null and alternative hypotheses are

- H<sub>0</sub>: there is no difference between treatment groups;
- H<sub>a</sub>: there is a difference between treatment groups.

While for this proof of concept study statistical significance (p<0.05) may not be achieved, these results will drive sample size projections for future studies. Due to the exploratory nature of the study, no adjustment to the alpha level for multiple comparisons will be made. P-values resulting from inferential testing will be considered primarily as summary statistics.

No statistical comparisons between the positive control regimen and the test product regimen are planned. The positive control is included to provide internal validation to the trial and to provide a reference point for estimates of effect size.

#### 4.4.1 Primary Efficacy Endpoint

#### 4.4.1.1 Primary Efficacy Endpoint Definition

The corneometer measurement of each subject at each assessment point will be calculated as the mean of the three repeated measurements of the subject at that assessment point.

The primary endpoint is the change from baseline in Corneometer measurement at 8 hours following the first product application. Data for the endpoint will be summarized by age stratum and treatment regimen (Table 14.2.2.2, 14.2.2.3 for the ITT population and Table 14.2.2.5, 14.2.2.6 for the PP population).

#### 4.4.1.2 Statistical Hypothesis, Model, and Method of Analysis

Analysis of covariance (ANCOVA) will be applied with treatment as main effect, age stratification and baseline measurement as covariate. Least squares means and differences between least squares means for (i) test product and no treatment regimen; (ii) positive control and no treatment regimen will be presented, together with 95% confidence intervals (Table 14.2.2.1 for the ITT population, Table 14.2.2.4 for the PP population).

In the randomisation stage of the study, a substantial number of subjects were randomised using wrong age stratum randomisation scheme. In all summary and analyses involving age stratum, subjects will be assigned to correct age strata using their actual ages.

#### 4.4.1.3 Supportive Analyses

The normality assumption for ANCOVA in primary analysis will be checked. If violated, non-parametric method such as Wilcoxon rank sum test may be applied.

#### 4.4.2 Secondary Efficacy Variables

Secondary efficacy variables of the study are listed below.

#### 4.4.2.1 Corneometer measurements at other time points

The change from baseline in Corneometer measurements at 1 and 3 hours following the first product application as well as at Weeks 1, 4 and 8 are secondary variables which will be summarized by age strata, treatment regimen and study visit (Table 14.2.2.2, 14.2.2.3 for the ITT population and Table 14.2.1.5, 14.2.1.6 for the PP population).

#### 4.4.2.2 Sebumeter and sebum excretion rate

The sebumeter measurement of each subject at each visit will be calculated as the mean of the three repeated assessments of the subject at that visit. The sebum excretion rate of each subject at each visit will be calculated as the difference of sebumeter kinetic measurement 90 mins post forehead cleansing to 5 mins post forehead cleansing. The sebumetry and sebum excretion rate changes from baseline at Weeks 1, 4 and 8 are secondary variables which will be summarized by age strata, treatment regimen and study visit (Table 14.2.3.2, 14.2.3.3 for sebumeter and Table 14.2.4.2, 14.2.4.3 for sebum excretion rate, ITT population).

#### 4.4.2.3 Blemish counts

Clinical assessment of blemish counts (papules and pustules) change from baseline at Weeks 1, 4 and 8 are secondary variables which will be summarized by age stratum, treatment regimen and study visit (Table 14.2.5.2, 14.2.5.3 for the ITT population and Table 14.2.5.5, 14.2.5.6 for the PP population).

#### 4.4.2.4 Lay person assessment

The lay person assessment resulting from the ranking of blemish images (Week 8 image vs. Baseline image with judgement either 'Week 8 is better' or 'Baseline is better') is a secondary variable. The assessment will be performed using polarised images and non-polarised images separately by 24 raters. Summary statistics will be provided by treatment (Table 14.2.6.2, for polarized image, Table 14.2.7.2 for non-polarised image, ITT population).

#### 4.4.3 Handling of Missing Values/Censoring/Discontinuations

Missing data will not be replaced or imputed. Dropouts will be included in analyses up to the point of discontinuation.

#### 4.5 Analysis of Secondary Objectives

#### 4.5.1 Efficacy

The change from baseline in corneometer measurements at 1 and 3 hours following the first product application as well as at Weeks 1, 4 and 8 will be analysed at each post-baseline time point using the same ANCOVA model as in primary analysis. Differences between least squares means for (i) test product and no treatment regimen; (ii) positive control and no treatment regimen will be presented, together with 95% confidence intervals. The normality assumption for ANCOVA will be checked. If violated, non-parametric method such as Wilcoxon rank sum test may be applied.

The sebumeter and sebumeter excretion rate changes from baseline at Weeks 1, 4 and 8 will be analysed at each post-baseline visit using ANCOVA with treatment main effect, age stratum (<21, ≥21 years of age) and baseline count as covariate. Differences between least squares means for (i) test product and no treatment regimen; (ii) positive control and no treatment regimen will be presented, together with 95% confidence intervals (Table 14.2.3.1 for sebumeter, Table 14.2.4.1 for sebumeter excretion rate). The normality assumption for ANCOVA will be checked. If violated, non-parametric method such as Wilcoxon rank sum test may be applied.

Clinical assessment of blemish counts (papules and pustules) change from baseline at Weeks 1, 4 and 8 will be analysed at each post-baseline visit using ANCOVA with treatment main effect, age stratum (<21, ≥21 years of age) and baseline count as covariate. Differences between least squares means for (i) test product and no treatment regimen; (ii) positive control and no treatment regimen will be presented, together with 95% confidence intervals (Table 14.2.5.1 for the ITT population and Table 14.2.5.4 for the PP population). The normality assumption for ANCOVA will be checked. If violated, non-parametric method such as Wilcoxon rank sum test may be applied. A figure will be provided for blemish profile of the ITT population (Figure 14.2.1).

The summary and analysis of lay person image assessment will be performed for polarised images and non-polarised images separately. Proportion of subjects evaluated as 'Week 8 is better' will be tabulated by treatment group and rater. Data from all 24 raters will also be pooled and a repeated measure logistic regression will be applied including effects of treatment and age stratum and exchangeable correlation structure among repeats. Odds ratio between (i) test product and no treatment regimen; (ii) positive control and no treatment regimen will be provided together with its 95%CI (Table 14.2.6.1 for polarised image, Table

14.2.7.1 for non-polarised image). This analysis will not be performed if all subjects are judged by all raters as 'Week 8 is better'.

#### 4.5.2 Pharmacokinetic (Secondary)

Not applicable.

#### 4.6 Analysis of Safety

#### 4.6.1 Adverse Events and Serious Adverse Events

All adverse events (AEs) will be summarised by system organ class and preferred term.

Treatment emergent adverse events (TEAEs), defined as the AEs reported after study product application (for the untreated group, TEAE is defined as first application of the standard cleanser), will be summarized by treatment and overall including the number and percentage of subjects having AEs and total number of AEs in each SOC and preferred term (Table 14.3.1.1). TEAEs will also be tabulated by severity (Table 14.3.1.2). Treatment-related TEAEs will be summarized and presented in the same manner (Table 14.3.1.3, Table 14.3.1.4).

Deaths occurring during treatment (if any) will be listed (Listing 14.3.2.1) by treatment, including the date and study day of death, and the principal cause of death. Non-fatal serious adverse events and TEAEs causing study treatment discontinuation will be listed (Listing 14.3.2.2, 14.3.2.3).

All AEs will be listed in the Listing 16.2.7.1 for randomised subjects and Listing 16.2.7.2 for non-randomised subjects.

#### 4.6.2 Other Safety Variables

Not applicable.

#### 4.7 Analysis of Other Variables

Not applicable.

#### 5 Changes to the Protocol Defined Statistical Analysis Plan

Any changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis section | Statistical Analysis Plan | Rationale for Changes |
| Section 9.3.2 and Section 9.3.3 | Section 2.4.1.2 and<br>Section 2.5 | Protocol analysis sections (9.3.2 and 9.3.3) mentions only the comparison between test product and no treatment regimen. In this SAP (Section 2.4.1.2 and Section 2.5) comparison between positive control and no treatment regimen is also included as required by client. |
| • Section 9.3.3 | • Section 2.5 | Protocol analysis section (9.3.3) states the blemish counts will be summarized and compared between treatment groups. This has been changed in Section 2.5 of the SAP to blemish change from baseline as required by client. |

## **Attachment 1: List of Data Displays**



#### **Attachment 2: Template for Tables, Figures and Listings**

This is a guideline which will give the guidance of treatment labels that will be used for the table header and in the figures, listings and in the footnotes.

The treatment labels for the column heading will be as follow:

- Test Product
- Untreated
- Positive Control



Protocol 207196

Table 14.1.1
Subject Disposition
All Screened Subjects

Program Run Date:xxxx

All Screened Subjects (N=xxx)

| | Test Product | Untreated | Positive Control | Overall |
|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) |
| TOTAL SUBJECTS SCREENED | | | | xxx |
| TOTAL SUBSCISS SCIENCE | | | | ^^^ |
| SUBJECTS NOT RANDOMISED | | | | Xxx (xx.x) |
| DID NOT MEET STUDY CRITERIA | | | | xxx (xx.x) |
| ADVERSE EVENT | | | | Xxx (xx.x) |
| LOST TO FOLLOW UP | | | | xxx (xx.x) |
| PROTOCOL VIOLATION | | | | Xxx (xx.x) |
| WITHDRAWAL OF CONSENT | | | | Xxx (xx.x) |
| OTHER | | | | Xxx (xx.x) |
| SUBJECTS RANDOMISED | xxx | xxx | xxx | Xxx |
| COMPLETED STUDY | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DID NOT COMPLETE STUDY | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DID NOT MEET STUDY CRITERIA | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ADVERSE EVENT | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| LOST TO FOLLOW-UP | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PROTOCOL VIOLATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WITHDRAWAL OF CONSENT | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| OTHER | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |




#### 207196

Statistical Reporting and Analysis plan, 19 Sep 2017

| | Test Product | Untreated | Positive Control | Overall |
|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) |
| SAFETY POPULATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ITT POPULATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PP POPULATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Page x of y

#### PPD

Programming note: For categories under 'Subjects Not Randomised' percentages will be calculated using the number of 'All Screened Subjects' as the denominator. Percentages under the 'Subjects Randomised' categories will be computed using number of subjects randomised as the denominator.



Protocol 207196 Program Run Date:xxxx

# Table 14.1.2 Incidence of Major Protocol Deviations Randomised Population

Intent-to-Treat Population (N=xxx)

| | Test Product<br>N (%) | Untreated<br>N (%) | Positive Control<br>N (%) | Overall<br>N (%) |
|---|---|---|---|---|
| NUMBER OF SUBJECTS WITH AT LEAST ONE MAJOR PROTOCOL VIOLATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| VIOLATION 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| VIOLATION 2 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| VIOLATION 3 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| VIOLATION 4 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ••• | | | | |

Page x of y

PPD



Protocol 207196 Program Run Date:xxxx

Table 14.1.3 Analysis of Population Randomised Population

Intent-to-Treat Population (N=xxx)

| | Test Product<br>N (%) | Untreate<br>N ( | | ive Control<br>(%) | Overall<br>N (%) |
|---|---|---|---|---|---|
| NUMBER OF SUBJECTS EXCLUDED FROM SAFETY POPULATION | xxx (xx.x) | xxx (x | x.x) xxx | (xx.x) | xxx (xx.x) |
| DEVIATION 1 | xxx (xx.x) | • | - | (xx.x) | xxx (xx.x) |
| DEVIATION 2 | xxx (xx.x) | xxx (x | x.x) xxx | (xx.x) | xxx (xx.x) |
| NUMBER OF SUBJECTS EXCLUDED FROM ITT POPULATION | xxx (xx.x) | xxx (x | x.x) xxx | (xx.x) | xxx (xx.x) |
| DEVIATION 1 | xxx (xx.x) | xxx (x | x.x) xxx | (xx.x) | xxx (xx.x) |
| DEVIATION 2 | xxx (xx.x) | xxx (x | x.x) xxx | (xx.x) | xxx (xx.x) |
| ••• | | | | | |
| NUMBER OF SUBJECTS WITH AT LEAST ONE<br>DATA POINT EXCLUDED FROM PP ANALYSIS | | xxx (x | x.x) xxx | (xx.x) | xxx (xx.x) |
| NUMBER OF SUBJECTS EXCLUDED FROM PP POPULATION | xxx (xx.x) | xxx (x | x.x) xxx | (xx.x) | xxx (xx.x) |
| PROTOCOL VIOLATIONS LEADING TO EXCLUSION FROM PP | | | | | |
| All VISITS | | | | | |
| DEVIATION 1 | xxx (xx.x) | xxx (x | x.x) xxx | (xx.x) | xxx (xx.x) |
| DEVIATION 2 | xxx (xx.x) | xxx (x | x.x) xxx | (xx.x) | xxx (xx.x) |




#### 207196

#### Statistical Reporting and Analysis plan, 19 Sep 2017

| | Test Product<br>N (%) | Untreated<br>N (%) | Positive Control<br>N (%) | Overall<br>N (%) |
|---|---|---|---|---|
| • • • | | | | |
| ISIT3 / WEEK2 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DEVIATION 3 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DEVIATION 4 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ••• | | | | |
| ISIT4 / WEEK4 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DEVIATION 5 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DEVIATION 6 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Page x of y

PPD



Protocol 207196 Program Run Date:xxxx

# Table 14.1.4.1 Subject Demographics and Baseline Characteristics Safety Population

Safety Population (N=XX)

| covery repulses with the control of | Test Product<br>(N=XX) | Untreated<br>(N=XX) | Positive Control<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| SEX n (%) | | | | |
| MALE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| FEMALE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| RACE n (%) | | | | |
| ASIAN | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AFRICAN AMERICAN | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AMERICAN INDIAN OR ALASKA NATIVE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| WHITE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| (as in eCRF) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AGE (YEARS) | | | | |
| n | XX | XX | xx | XX |
| MEAN | XX.X | XX.X | xx.x | XX.X |
| SD | XX.XX | XX.XX | xx.xx | XX.XX |
| MEDIAN | XX.X | XX.X | xx.x | XX.X |
| MINIMUM | XX | XX | XX | XX |



#### 207196

#### Statistical Reporting and Analysis plan, 19 Sep 2017

| | Test Product<br>(N=XX) | Untreated<br>(N=XX) | Positive Control<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| MAXIMUM | XX | XX | XX | XX |
| FITZPATRICK SCALE FOR SKIN 1 | ТҮРЕ | | | |
| I | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| II | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| III | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| IV | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| V | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| VI | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AGE STRATA (By Planned Rando | omisation) | | | |
| Age < 21 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Age ≥ 21 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AGE STRATA (By Actual Age) | | | | |
| Age < 21 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Age ≥ 21 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Fitzpatrick Scale I: Always burns, never tans II: Usually burns, tans minimally III: Sometimes mild burn, tans uniformly (cream white; fair with any hair or eye color) IV: Burns minimally, always tans well (moderate brown) V: very rarely burns, tans very easily (dark brown). VI Never burns, never tans (deeply pigmented dark brown to darkest brown).

Page x of y

PPD



#### 207196

#### Statistical Reporting and Analysis plan, 19 Sep 2017

Protocol 207196 Program Run Date:xxxx

#### Table 14.2.1 Compliance\* Intent-to-Treat Population

Intent-to-Treat Population(N=XX)

| Compliance<br>Period | Product | Test product (N=XX) | Untreated (N=XX) | Positive Control (N=XX) |
|---|---|---|---|---|
| V2 to V3 | Cream<br>Cleanser | MEAN (SD) Median (MIN, MAX) x.xx(x.xxx) x.xx(x.xx, x.xx) x.xx(x.xxx) x.xx(x.xx, x.xx) | MEAN (SD) Median (MIN, MAX) x.xx(x.xxx) x.xx(x.xx, x.xx) | MEAN (SD) Median (MIN, MAX) x.xx(x.xxx) x.xx(x.xx, x.xx) x.xx(x.xxx) x.xx(x.xx, x.xx) |
| V3 to V4 | Cream<br>Cleanser | | | |
| V4 to V5 | Cream<br>Cleanser | | | |

<sup>\*</sup>Compliance = Actual Number of Uses / Expected Number of Uses

Page x of y

PPD

Programming Note: For each subject, Total Expected = 2\*Number of Days Between the Two Visits; Actual Uses = Expected Number - Missed Uses + Extra Uses. For untreated group, only cleasner row to be filled.



Program Run Date:xxxx Protocol 207196

#### Table 14.2.2.1 Analysis of Corneometer Change from Baseline Intent-to-Treat Population

| Intent-to-Treat Popula | ation( | (N=XX) |
|------------------------|--------|--------|
|------------------------|--------|--------|

| Visit | | Variable | Test Product | Untreated | Positive Control |
|---|---|---|---|---|---|
| | | | (N=XX) | (N=XX) | (N=XX) |
| 1 Hour Change from<br>Baseline | | | | | |
| | | LSmeans(SE), p-value[1] | X.xx(x.xxx), 0.xxxx | X.xx(x.xxx), 0.xxxx | X.xx (x.xxx), 0.xxxx |
| | | Comparison[1][2] | Difference | 95%CI | P-value |
| | | Test vs Untreat | x.xx | (x.xx, x.xx) | 0.xxxx |
| | | Positive v Untreat | x.xx | (x.xx, x.xx) | 0.xxxx |
| 3 Hours Change from<br>Baseline | (same template) | | | | |
| 8 Hours Change from<br>Baseline | (Same template) | | | | |
| 1 Week Change from<br>Baseline | (Same template) | | | | |
| 4 Week Change from<br>Baseline | (Same template) | | | | |
| 8 Week Change from<br>Baseline | (Same template) | | | | |

<sup>[1]</sup> From ANCOVA with treatment main effect, age stratum and baseline as covariate



[2] Difference is first named treatment minus second named treatment such that a negative difference favours the first named treatment

Page x of y

#### PPD

Programming Note: If non-parametric method is used due to the failure in ANCOVA model check, the following non-parametric results should be added to the table

| Comparison | P-value (Wilcoxon) |
|---------------------|--------------------|
| Test vs. Untreat | A 2000 |
| Positive vs Untreat | 0.xxxx<br>0.xxxx |



Protocol 207196 Program Run Date:xxxx

Table 14.2.2.2

Summary of Corneometer Change from Baseline
Intent-to-Treat Population

Intent-to-Treat Population(N=XX)

| Visit | Variable | Test Product | Untreated | Positive Control |
|---|---|---|---|---|
| | | (N=XX) | (N=XX) | (N=XX) |
| Baseline | n | Xx | Xx | Xx |
| | MEAN | x.xx | x.xx | x.xx |
| | SD | x.xxx | x.xxx | x.xxx |
| | MEDIAN | x.xx | x.xx | x.xx |
| | MINIMUM | X.xx | X.xx | X.xx |
| | MAXIMUM | X.xx | X.xx | X.xx |
| 1 Hour | | | | |
| | n | Xx | Xx | Xx |
| | MEAN | x.xx | x.xx | x.xx |
| | SD | x.xxx | x.xxx | x.xxx |
| | MEDIAN | x.x | x.x | x.x |
| | MINIMUM | X.x | X.x | X.x |
| | MAXIMUM | X.x | X.x | X.x |
| 1 Hour Change from<br>Baseline | | | | |
| | n | Xx | Xx | Xx |
| | MEAN | x.xx | x.xx | x.xx |
| | SD | x.xxx | x.xxx | x.xxx |

GlaxoSmithKline Consumer Healthcare Confidential

#### CC

#### 207196

#### Statistical Reporting and Analysis plan, 19 Sep 2017

| Visit | | Variable | Test Product | Untreated | Positive Control |
|---|---|---|---|---|---|
| | | | (N=XX) | (N=XX) | (N=XX) |
| | | MEDIAN | x.x | x.x | x.x |
| | | MINIMUM | X. x | X.x | X.x |
| | | MAXIMUM | X.x | X.x | X.x |
| 3 Hours | (same template) | | | | |
| 3 Hours Change from Baseline | (same template) | | | | |
| 8 Hours | (same template) | | | | |
| 8 Hours Change from<br>Baseline | (Same template) | | | | |
| 1 Week | (Same template) | | | | |
| 1 Week Change from<br>Baseline | (Same template) | | | | |
| 4 Week | (Same template) | | | | |
| 4 Week Change from<br>Baseline | (Same template) | | | | |
| 8 Week | (Same template) | | | | |
| 8 Week Change from<br>Baseline | (Same template) | | | | |

Page x of y

PPD



Protocol 207196 Program Run Date:xxxx

Table 14.2.2.3

Summary of Corneometer Change from Baseline by Age Strata
Intent-to-Treat Population

Intent-to-Treat Population (N=XX)

| Visit | Stratum | Variable | Test Product | Untreated (N=XX) | Positive Control (N=XX) |
|---|---|---|---|---|---|
| | | | (N=XX) | | |
| Baseline | Age<21 | n | Xx | Xx | Xx |
| | | MEAN | x.xx | x.xx | x.xx |
| | | SD | x.xxx | x.xxx | x.xxx |
| | | MEDIAN | x.xx | x.xx | x.xx |
| | | MINIMUM | X.xx | X.xx | X.xx |
| | | MAXIMUM | X.xx | X.xx | X.xx |
| | Age≥21 | n | Xx | Xx | Xx |
| | | MEAN | x.xx | x.xx | x.xx |
| | | SD | x.xxx | x.xxx | x.xxx |
| | | MEDIAN | x.xx | x.xx | x.xx |
| | | MINIMUM | X.xx | X.xx | X.xx |
| | | MAXIMUM | X.xx | X.xx | X.xx |
| 1 Hour | Age<21 | n | Xx | Xx | Xx |
| 1 11041 | Thou | MEAN | x.xx | x.xx | x.xx |
| | | SD | x.xxx | x.xxx | x.xxx |
| | | MEDIAN | x.xx | x.xx | x.xx |
| | | MINIMUM | X.xx | X.xx | X.xx |

**CCI** 207196

| Visit | Stratum | Variable | Test Product | Untreated (N=XX) | Positive Control (N=XX) |
|---|---|---|---|---|---|
| | | | (N=XX) | | |
| | | MAXIMUM | X.xx | X.xx | X.xx |
| | Age≥21 | n | Xx | Xx | Xx |
| | | MEAN | x.xx | x.xx | x.xx |
| | | SD | x.xxx | x.xxx | x.xxx |
| | | MEDIAN | x.xx | x.xx | x.xx |
| | | MINIMUM | X.xx | X.xx | X.xx |
| | | MAXIMUM | X.xx | X.xx | X.xx |
| 1 Hour Change from Age<<br>Baseline | Age<21 | n | Xx | Xx | Xx |
| | | MEAN | x.xx | x.xx | x.xx |
| | | SD | x.xxx | x.xxx | x.xxx |
| | | MEDIAN | x.xx | x.xx | x.xx |
| | | MINIMUM | X.xx | X.xx | X.xx |
| | | MAXIMUM | X.xx | X.xx | X.xx |
| | Age≥21 | n | Xx | Xx | Xx |
| | | MEAN | x.xx | x.xx | x.xx |
| | | SD | x.xxx | x.xxx | x.xxx |
| | | MEDIAN | x.xx | x.xx | x.xx |
| | | MINIMUM | X.xx | X.xx | X.xx |
| | | MAXIMUM | X.xx | X.xx | X.xx |
| Hour | (same templa | te) | | | |
| Hours Change from | (Same templa | te) | | | |

#### CCI

#### 207196

#### Statistical Reporting and Analysis plan, 19 Sep 2017

| Visit | Stratum | Variable | Test Product | Untreated (N=XX) | Positive Control (N=XX) |
|---|---|---|---|---|---|
| | | | (N=XX) | | |
| Baseline | | | | | |
| 8 Hour | (same template) | | | | |
| 8 Hours Change from<br>Baseline | (Same template) | | | | |
| 1 Week | (Same template) | | | | |
| 1 Week Change from<br>Baseline | (Same template) | | | | |
| 4 Week | (Same template) | | | | |
| 4 Week Change from<br>Baseline | (Same template) | | | | |
| 8 Week | | | | | |
| 8 Week Change from<br>Baseline | (Same template) | | | | |

PPD

Page x of y


Protocol 207196 Program Run Date:xxxx

## Table 14.2.3.1 Analysis of Sebumeter Change from Baseline Intent-to-Treat Population

#### Intent-to-Treat Population(N=XX)

| Visit | | Variable | Test Product | Untreated (N=XX) | Positive Control (N=XX) |
|---|---|---|---|---|---|
| | | | (N=XX) | | |
| 1 Week Change from<br>Baseline | | | | | |
| | | LSmeans(SE), p-value | X.xx (x.xxx), 0.xxxx | X.xx (x.xxx), 0.xxxx | X.xx (x.xxx), 0.xxxx |
| | | Comparison[1][2] | Difference | 95%CI | P-value |
| | | Test vs Untreat | x.xx | (x.xx, x.xx) | 0.xxxx |
| | | Positive vs Untreat | x.xx | (x.xx, x.xx) | 0.xxxx |
| 4 Week Change from<br>Baseline | (same template) | | | | |
| 8 Week Change from<br>Baseline | (Same template) | | | | |

- [1] From ANCOVA with treatment main effect, age stratum and baseline as covariate
- [2] Difference is first named treatment minus second named treatment such that a negative difference favours the first named treatment

Page x of y



Protocol 207196 Program Run Date:xxxx

## Table 14.2.3.2 Summary of Sebumeter Change from Baseline Intent-to-Treat Population

#### Intent-to-Treat Population(N=XX)

| Visit | Variable | Test Product | Untreated (N=XX) | Positive Control (N=XX) |
|---|---|---|---|---|
| | | (N=XX) | | |
| Baseline | n | Xx | Xx | Xx |
| | MEAN | x.xx | x.xx | x.xx |
| | SD | x.xxx | x.xxx | x.xxx |
| | MEDIAN | x.xx | x.xx | x.xx |
| | MINIMUM | X.xx | X.xx | X.xx |
| | MAXIMUM | X.xx | X.xx | X.xx |
| 1 Week | n | Xx | Xx | Xx |
| | MEAN | x.xx | x.xx | x.xx |
| | SD | x.xxx | x.xxx | x.xxx |
| | MEDIAN | x.xx | x.xx | x.xx |
| | MINIMUM | X.xx | X.xx | X.xx |
| | MAXIMUM | X.xx | X.xx | X.xx |
| 1 Week Change from | n | Xx | Xx | Xx |
| Baseline | | | | |
| | MEAN | x.xx | x.xx | x.xx |
| | SD | x.xxx | x.xxx | x.xxx |
| | MEDIAN | x.x | x.x | x.x |




### 207196

### Statistical Reporting and Analysis plan, 19 Sep 2017

| Visit | | Variable | Test Product | Untreated (N=XX) | Positive Control (N=XX) |
|---|---|---|---|---|---|
| | | | (N=XX) | | |
| | | MINIMUM | X.x | X.x | X.x |
| | | MAXIMUM | X.x | X.x | X.x |
| 4 Week 4 Week Change from | <pre>(same template) (Same template)</pre> | | | | |
| Baseline | (Same template) | | | | |
| 8 Week | (Same template) | | | | |
| 8 Week Change from<br>Baseline | (Same template) | | | | |

Page x of y



Protocol 207196 Program Run Date:xxxx

Table 14.2.3.3

Summary of Sebumeter Change from Baseline by Age Strata
Intent-to-Treat Population

Intent-to-Treat Population(N=XX)

| Visit | Stratum | Variable | Test Product | Untreated | Positive Control (N=XX) |
|---|---|---|---|---|---|
| | | | (N=XX) | (N=XX) | |
| Baseline | Age<21 | n | Xx | Xx | Xx |
| | | MEAN | x.xx | x.xx | x.xx |
| | | SD | x.xxx | x.xxx | x.xxx |
| | | MEDIAN | x.xx | x.xx | x.xx |
| | | MINIMUM | X.xx | X.xx | X.xx |
| | | MAXIMUM | X.xx | X.xx | X.xx |
| | Age≥21 | n | Xx | Xx | Xx |
| | | MEAN | x.xx | x.xx | x.xx |
| | | SD | x.xxx | x.xxx | x.xxx |
| | | MEDIAN | x.xx | x.xx | x.xx |
| | | MINIMUM | X.xx | X.xx | X.xx |
| | | MAXIMUM | X.xx | X.xx | X.xx |
| 1 Week | Age<21 | n | Xx | Xx | Xx |
| 1 Neek | | MEAN | x.xx | x.xx | x.xx |
| | | SD | x.xxx | x.xxx | x.xxx |
| | | MEDIAN | x.xx | x.xx | x.xx |
| | | MINIMUM | X.xx | X.xx | X.xx |

CCI 207196

| Visit | Stratum | Variable | Test Product | Untreated | Positive Control (N=XX) |
|---|---|---|---|---|---|
| | | | (N=XX) | (N=XX) | |
| | | MAXIMUM | X.xx | X.xx | X.xx |
| | Age≥21 | n | Xx | Xx | Xx |
| | | MEAN | x.xx | x.xx | x.xx |
| | | SD | x.xxx | x.xxx | x.xxx |
| | | MEDIAN | x.xx | x.xx | x.xx |
| | | MINIMUM | X.xx | X.xx | X.xx |
| | | MAXIMUM | X.xx | X.xx | X.xx |
| 1 Week Change from<br>Baseline | | | | | |
| | Age<21 | n | Xx | Xx | Xx |
| | | MEAN | x.xx | x.xx | x.xx |
| | | SD | x.xxx | x.xxx | x.xxx |
| | | MEDIAN | x.xx | x.xx | x.xx |
| | | MINIMUM | X.xx | X.xx | X.xx |
| | | MAXIMUM | X.xx | X.xx | X.xx |
| | Age≥21 | n | Xx | Xx | Xx |
| | | MEAN | x.xx | x.xx | x.xx |
| | | SD | x.xxx | x.xxx | x.xxx |
| | | MEDIAN | x.xx | x.xx | x.xx |
| | | MINIMUM | X.xx | X.xx | X.xx |
| | | MAXIMUM | X.xx | X.xx | X.xx |
| 4 Week | (Same templat | e) | | | |



### 207196

### Statistical Reporting and Analysis plan, 19 Sep 2017

| Visit | Stratum | Variable | Test Product | Untreated | Positive Control (N=XX) |
|---|---|---|---|---|---|
| | | | (N=XX) | (N=XX) | |
| 4 Week Change from<br>Baseline | (Same template) | | | | |
| 8 Week | (Same template) | | | | |
| 8 Week Change from<br>Baseline | (Same template) | | | | |

PPD

Page x of y



Protocol 207196 Program Run Date:xxxx

# Table 14.2.6.1 Analysis of Lay Person Assessment Polarised Image Intent-to-Treat Population

#### Intent-to-Treat Population(N=XX)

| Variable | Test Product | Untreated (N=XX) | Positive Control (N=XX) |
|------------------|--------------|------------------|-------------------------|
| | (N=XX) | | |
| ODDS[1] | xx.xx | Xx.xx | Xx.xx |
| Comparison[1][2] | ODDS RATIO | 95%CI | p-value |
| Test vs. Control | xx.xx | (xx.xx, xx.xx) | 0.xxxx |

ODDS=p/(1-p) where p is the probability of event that week 8 is better than baseline.

- [1] From logistic regression including treatment and age stratum effects and exchangeable correlation structure among repeats
- [2] Odds ratio is the first named treatment over the second named treatment such that ratio > 1 favours the first named treatment

Page x of y



Protocol 207196 Program Run Date:xxxx

## Table 14.2.6.2 Summary of Lay Person Assessment Polarised Image by Rater Intent-to-Treat Population

#### Intent-to-Treat Population(N=XX)

| Rater | Number of Subjects | Variable | Test Product | Untreated | |
|---|---|---|---|---|---|
| | Assessed | | (N=XX) | (N=XX) | Positive Control (N=XX) |
| 01 | xx | Proportion<br>(Week 8 is better) | Xx . x% | Xx.x% | Xx.x% |
| 02 | xx | Proportion<br>(Week 8 is better) | Xx . x% | Xx.x% | Xx.x% |
| ••• | | | | | |
| 24 | xx | Proportion<br>(Week 8 is better) | Xx.x% | Xx.x% | Xx.x% |

Page x of y



#### 207196

#### Statistical Reporting and Analysis plan, 19 Sep 2017

Protocol 207196 Program Run Date:xxxx

Table 14.3.1.1

Treatment Emergent Adverse Event by System Organ Class and Preferred Term
Safety Population

| | | | barce, reputation | | | |
|---|---|---|---|---|---|---|
| Safety Population (N=xx) | | | | | | |
| System Organ Class<br>Preferred Term | Test Pro | duct | Untreated (N=XX) | | Overal | .1 |
| Preferred Term | | | (, | | | |
| | (N=X | X) | | Positive Control (N=xx) | (N=XX) | ) |
| <del>-</del> | n (%) | nAE | | | n (%) | nAE |
| UMBER OF SUBJECTS WITH AT | xx (xx.x) | xx | | | xx (xx.x) | xx |
| NUMBER OF SUBJECTS WITH NO<br>FEAE | xx (xx.x) | xx | | | xx (xx.x) | xx |
| KIN AND SUBCUTANEOUS | xx (xx.x) | xx | | | xx (xx.x) | xx |
| ERYTHEMA | xx (xx.x) | XX | | | xx (xx.x) | xx |
| DERMATITIS | xx (xx.x) | xx | • | ••• | xx (xx.x) | XX |
| GASTROINTESTINAL SYSTEM | xx (xx.x) | xx | | | xx (xx.x) | xx |
| ABDOMINAL PAIN | xx (xx.x) | xx | | | xx (xx.x) | xx |
| DRY MOUTH | xx (xx.x) | xx | | | xx (xx.x) | xx |
| VOMITTING | xx (xx.x) | XX | | | xx (xx.x) | xx |

n (%) = Number (percent) of subjects nAE = Number of adverse events.

Page x of y



Protocol 207196 Program Run Date:xxxx

Table 14.3.1.2

Treatment Emergent Adverse Event by System Organ Class, Preferred Term and Severity Safety Population

Safety Population (N=xx)

System Organ Class
Preferred Term

Test Product

(N=XX)

...

(N=XX)

| | Mild | | Moderat | te | Severe | 9 | | Mild | | Moderat | e | Severe | e |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | n (%) | nAE | n (%) | nAE | n (%) | nAE | | n (%) | nAE | n (%) | nAE | n (%) | nAE |
| NUMBER OF SUBJECTS | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| WITH AT LEAST ONE TEAE | | | | | | | | | | | | | |
| | | XX | | XX | | XX | | | XX | | XX | | XX |
| SKIN AND SUBCUTANEOUS | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | | xx(xx.x) | XX | xx(xx.x) | XX | xx (xx.x) | XX |
| TISSUE DISORDERS | | | | | | | | | | | | | |
| ERYTHEMA | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| DERMATITIS | xx (xx.x) | xx | xx (xx.x) | XX | xx (xx.x) | xx | • • • | xx (xx.x) | xx | xx (xx.x) | XX | xx (xx.x) | XX |
| GASTROINTESTINAL<br>SYSTEM | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | ••• | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| ABDOMINAL PAIN | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | | xx (xx.x) | xx | xx(xx.x) | XX | xx (xx.x) | XX |
| DRY MOUTH | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| VOMITTING | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |

n (%) = Number (percent) of subjects nAE = Number of adverse events.

Page x of y



Protocol 207196 Program Run Date:xxxx

Figure 14.2.1

Total Blemish Count Mean (±SE) Plot Over Time by Treatment
Intent-to-Treat Population

Intent-to-Treat Population (N=XX)



<sup>\*</sup> Significant change from baseline within group (p<0.05)

Page x of y

<sup>\*</sup> Significant treatment difference on change from baseline as compared to untreated (p<0.05)



Protocol 207196 Program Run Date:xxxx

# Listing 16.1.7 Randomisation Information Randomised Population

Stratum 1: Age<21

Subject Number Age/Sex/Race[1] Randomisation Number Treatment Randomised Date of Randomisation

PPD 32/F/W PPD 20-Mar-2017

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, O = Multiple.

Page x of y



Protocol 207196 Program Run Date:xxxx

Listing 16.2.1.1 Subject Disposition Randomised Population

Treatment Group: Test Product

| Subject | Age/Sex/ Race [1] | Screening<br>date | Treatment<br>Start Date<br>and Time | Date of<br>Completion or<br>withdrawal | Duration of<br>Treatment<br>(Days) | Completed<br>(Yes/No) | Primary Reason for<br>Withdrawal |
|---|---|---|---|---|---|---|---|
| PPD | | | | | | | |

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.

Page x of y

| CCI |
|--------|
| 207196 |

Protocol 207196 Program Run Date:xxxx

Listing 16.2.1.2 Subject Disposition Non-Randomised Subjects

| Subject<br>Number | Age/Sex/ Race [1] | Screening date | Reason of Screen failure |
|---|---|---|---|
| PPD | | | |

Page x of y

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.



Protocol 207196 Program Run Date:xxxx

Listing 16.2.2.1
Major Protocol Deviations
All Randomized Subjects

Treatment Group: XXXXXX

Week(s)/Time(s) Excluded from PP

Subject Sex/Age/ Race [1] Population Deviation Reason

#### PPD

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.

Page x of y



Protocol 207196 Program Run Date:xxxx

Listing 16.2.2.2 Minor Protocol Deviation Randomised Population

| PPD | | | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
|---|---|---|---|---|
| Number | Age/Sex/Race[1] | VISIC | Deviation Sequence | Protocol peviation |
| Subject | Age/Sex/Race[1] | Vi ci+ | Deviation Sequence | Protocol Deviation |
| Treatment ( | roup: Test Product | | | |

Page x of y

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, O = Multiple.



Protocol 207196 Program Run Date:xxxx

# Listing 16.2.3.1 Exclusions from Analysis Populations Randomised Population

| Treatment | Group: Test Product | | | | | |
|---|---|---|---|---|---|---|
| Subject | Age/Sex/Race[1] | Treatment Start Date | Safety Population | ITT Population | PP population | |
| Number | | and Time | (Yes/No) | (Yes/No) | (Yes/No) | |
| PPD | | | | | | _ |

Page x of y

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, O = Multiple.



Program Run Date:xxxx Protocol 207196

> Listing 16.2.4.1 Demographic Characteristics Randomised Population

Treatment Group: Test Product Fitzpatrick Skin Type Stratum (Actual) Subject Age Sex Race Stratum (Planned) Number (years)

Page x of y



Protocol 207196 Program Run Date:xxxx

## Listing 16.2.4.2 Medical History and Current Medical Conditions Randomised Population

Randomised Population

Treatment Group: Test Product

Age/Sex/Race Any Medical History?

Subject [1] (Yes/No) Medical Condition Start Date Ongoing? (Yes/No)

PPD

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.

Page x of y

End Date



Protocol 207196 Program Run Date:xxxx

## Listing 16.2.5.1 Study Product Administration and Compliance Randomised Population

Treatment Group: Test Product

Subject Age/Sex/Race[1] Administration (Yes/No) period Product Number Missed Extra

PPD

Number Missed Extra

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.

Page x of y



Protocol 207196 Program Run Date:xxxx

# Listing 16.2.5.2 Concomitant medications and significant non-drug therapies taken during treatment Randomised Population

| Treatment | droup: Test Produc | L | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Subject | Age/Sex/Race[1] | Sequence | Treatment | Reason of | Frequence | Start Date | Ongoing? (Yes/No) | End Date (Ongoing) |
| Number | | Number | | Treatment | | | | |
| PPD | | | | | | | | |

Page x of y

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.



Protocol 207196 Program Run Date:xxxx

Listing 16.2.6.1 Corneometer Measurement Randomised Population

Treatment Group: Test Product
Subject Age/Sex/Race[1] Visit Time Measurement 1 Measurement 2 Measurement 3 Mean Mean Change from Baseline
PPD

Page x of y

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.



Protocol 207196 Program Run Date:xxxx

## Listing 16.2.6.2 Sebumeter and Sebumeter Kinetic Measurements Randomised Population

| Treatment | Group: Test Product | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Age/Sex/Race[1] | Visit | Time | Measurement 1 | Measurement 2 | Measurement 3 | Mean | Mean Change from<br>baseline |
| PPD | | | | | | | | 22321110 |
| – | | | | | | | | |

Page x of y

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.



Protocol 207196 Program Run Date:xxxx

Listing 16.2.6.3

Blemish Count
Randomised Population

Treatment Group: Test Product

Subject Age/Sex/Race[1] Visit Papules Pustules Total Total Change from Number (Forehead, Cheeks, Chin) (Forehead, Cheeks, Chin) Baseline

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.

Page x of y



Protocol 207196 Program Run Date:xxxx

> Listing 16.2.6.4 Image assessment Randomised Population

Treatment Group: Test Product Age/Sex/Race[1] Subject Compare Image Score[2] Rater Number

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.

[2] Score: 0= Day1 image is better, 1= Day57 image is better.

Page x of y



Protocol 207196 Program Run Date:xxxx

Listing 16.2.7.1 All Adverse Events Randomised Population

Treatment Group: Test Product

| Subject | Age/Sex/ | Adverse | Start Date | Start | End Date | End | Frequ | Related to | Action | Outcome | Seri- | Withdrew? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Race[1] | Event (Preferred Term) (System | /Study<br>Day[2] | Time | | Time | ency<br>/Inte<br>nsity<br>[3] | Study<br>Product? | Taken re<br>Study<br>Product | | ous? | [4] |

PPD

Page x of y

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, O = Multiple.

<sup>[2]</sup> Study day is the day relative to start of treatment, day 1 being the day of first treatment.

<sup>[3]</sup> INT = Intermittent and SGLE = Single.

<sup>[4]</sup> Did subject withdraw from study as a result of this adverse event?



```
Programming Note for Listing 16.2.7.2:
Repeat the same layout for listing 16.2.7.2
Population should be used 'Non randomised Subjects'
The fourth column should be only 'Start Date'
Delete the footnote related to study day and adjust the numbers accordingly.
```



# STATISTICAL REPORTING AND ANALYSIS PLAN ADDENDUM 1

A randomised, parallel-group, evaluator-blind, no-treatment and positive controlled, single-site, proof of concept clinical study to evaluate the cosmetic benefit provided by 8 weeks of twice-daily topical application of a developmental moisturising cream with niacinamide in healthy subjects with sensitive, oily, blemish-prone skin

Protocol Number: 207196

Phase: NA

This document contains confidentiality statements that are not relevant for this publicly available version.

Property of GSK Consumer Healthcare
Confidential

May not be used, divulged, published or otherwise disclosed without the consent of GSK

Template Version Effective: 15-Jul-2017

Page 1 of 8

## **Document History**

| Document | Version Date | Summary of Changes (New analysis or Change in planned analysis) |
|---|---|---|
| Addendum 1 | 20-Dec-2017 | In addition to the planned analysis on lay rater image data as in RAP Section 4.5.1, an ANOVA on combined rate (over 24 raters) will be performed as requested by client. Table shell T 14.2.6.3 and T 14.2.7.3 are created for the ANOVA analysis of polarised image and non-polarised image respectively. |
| Original Analysis Plan | 19-Sept-2017 | Not applicable (N/A) |



### Statistical Reporting and Analysis plan Addendum 1, 20 Dec 2017

| Table of contents Document History | , |
|----------------------------------------|---|
| Table of contents | |
| 1 Introduction | |
| 4.5 Analysis of Secondary Objectives | 4 |
| 4.5.1 Efficacy | 4 |
| 5 Changes to Statistical Analysis Plan | 5 |
| Attachment Template for Table | |



#### 1 Introduction

This RAP addendum describes an analysis and its outputs in addition to those planned in the Statistical Reporting and Analysis Plan (V1.0, 19-Sept-2017) and Study protocol (V4.0, 23-May-2017). This analysis was requested by client after study unblinding but prior to final CSR. This additional analysis will be reported in the final CSR.

The sections below provide the updated text to that of the RAP Section 4.5 for the analyses of the secondary objectives, with Section 5.0 providing further details on what was planned, the additional and the reason for the additional. A summary of the additional analysis is as the following.

Lay person assessment of the appearance of blemishes was one of the secondary endpoints of the study. There were 24 raters and each gave a score 1 or 0 to each subject (indicating if Week 8 image was better than baseline image or not). An additional analysis on this endpoint was requested by client to average the 24 rating scores within a subject and then apply an ANOVA analysis to the average rates of all subjects including effects of treatment and age stratum.

### 4.5 Analysis of Secondary Objectives

#### 4.5.1 Efficacy

The summary and analysis of lay person image assessment will be performed for polarised images and non-polarised images separately. Proportion of subjects evaluated as 'Week 8 is better' will be tabulated by treatment group and rater. Data from all 24 raters will also be pooled and a repeated measure logistic regression will be applied including effects of treatment and age stratum and exchangeable correlation structure among repeats. Odds ratio between (i) test product and no treatment regimen; (ii) positive control and no treatment regimen will be provided together with its 95%CI (Table 14.2.6.1 for polarised image, Table 14.2.7.1 for non-polarised image). This analysis will not be performed if all subjects are judged by all raters as 'Week 8 is better'.

Here 'Week 8 is better' implies Week 8 shows less blemishes than baseline.

Data from all 24 raters for each subject will be combined into average rate - the mean of missing scores from 24 raters. An ANOVA analysis will then be applied with factors for treatment and age stratum. Mean treatment responses and differences between (i) test product and no treatment regimen; (ii) positive control and no treatment regimen will be provided together with 95%CIs (Table 14.2.6.3 for polarised image, Table 14.2.7.3 for non-polarised image, ITT population).



### 5 Changes to Statistical Analysis Plan

There is no change to the planned analysis in RAP (dated 19 Sept 2017). An additional analysis is added as outlined in Table 1.

Table 1 Additional to RAP Defined Analysis Plan

| Analysis in RAP | Additional in RAP addendum | Rationale for the additional |
|---|---|---|
| • Last Paragraph of Section 4.5.1 The summary and analysis of lay person image assessment will be performed for polarised images and non-polarised images separately. Proportion of subjects evaluated as 'Week 8 is better' will be tabulated by treatment group and rater. Data from all 24 raters will also be pooled and a repeated measure logistic regression will be applied including effects of treatment and age stratum and exchangeable correlation structure among repeats. Odds ratio between (i) test product and no treatment regimen; (ii) positive control and no treatment regimen will be provided together with its 95%CI (Table 14.2.6.1 for polarised image, Table 14.2.7.1 for non-polarised image). This analysis will not be performed if all subjects are judged by all raters as 'Week 8 is better' | • Last two Paragraphs of Section 4.5.1 The summary and analysis of lay person image assessment will be performed for polarised images and non-polarised images separately. Proportion of subjects evaluated as 'Week 8 is better' will be tabulated by treatment group and rater. Data from all 24 raters will also be pooled and a repeated measure logistic regression will be applied including effects of treatment and age stratum and exchangeable correlation structure among repeats. Odds ratio between (i) test product and no treatment regimen; (ii) positive control and no treatment regimen will be provided together with its 95%CI (Table 14.2.6.1 for polarised image, Table 14.2.7.1 for non-polarised image). This analysis will not be performed if all subjects are judged by all raters as 'Week 8 is better'. Here 'Week 8 is better' implies Week 8 shows less blemishes than baseline. Data from all 24 raters for each subject will be combined into average rate, An ANOVA analysis will then be applied including effects of treatment | GSKCH requested an additional analysis due to the following observations. (i) In the planned repeated measurement logistic analysis, correlation structure among repeated assessments could have different choices and the robustness of the results with respect to different choices of correlation was unsure. (ii) Treatment evaluation and treatment comparison in terms of odds and oddsratio in the planned analysis were not as intuitive as rate and rate difference. An alternative would be to remove the correlation by combining the 24 rating scores within a subject to get an average rating for the subject (equivalent to proportion of raters who rate W8 image of the subject better than the baseline image). |

### Statistical Reporting and Analysis plan Addendum 1, 20 Dec 2017

| Analysis in RAP | Additional in RAP addendum | Rationale for the additional |
|---|---|---|
| | and age stratum. Treatment | |
| | differences on average rate | |
| | between (i) test product and no | |
| | treatment regimen; (ii) positive | |
| | control and no treatment | |
| | regimen will be provided | |
| | together with its 95%Cl (Table | |
| | 14.2.6.3 for polarised image, | |
| | Table 14.2.7.3 for non-polarised | |
| | image_ITT population). | |

### Attachment Template for Table

Protocol 207196 Program Run Date:xxxx

#### Intent-to-Treat Population(N=XX)

| Visit | Variable | Test Product | Untreated | Positive Control |
|---|---|---|---|---|
| | | (N=XX) | (N=XX) | (N=XX) |
| Week 8 | LSmeans(SE)[1] | x.xx (x.xxx) | x.xx (x.xxx) | x.xx (x.xxx) |
| | Comparison[1][2] | Difference | 95%CI | p-value |
| | Test vs. Untreated | x.xx | (x.xx, x.xx) | 0.xxx |
| | Positive vs. Untreated | x.xx | (x.xx, x.xx) | 0.xxxx |

<sup>[1]</sup> From ANOVA on average rate over all raters including effects of treatment and age stratum.

Page x of y

CC

<sup>[2]</sup> Difference is the first named treatment minus the second named treatment such that a positive difference favours the first named treatment



### Statistical Reporting and Analysis plan Addendum 1, 13 Dec 2017

Protocol 207196 Program Run Date:xxxx

## Table 14.2.7.3 Analysis of Lay Person Assessment Combined Rating for Non-Polarised Image Intent-to-Treat Population

#### Intent-to-Treat Population(N=XX)

| Visit | Variable | Test Product | Untreated | Positive Control |
|---|---|---|---|---|
| | | (N=XX) | (N=XX) | (N=XX) |
| Week 8 | LSmeans(SE)[1] | x.xx (x.xxx) | x.xx (x.xxx) | x.xx (x.xxx) |
| | Comparison[1][2] | Difference | 95%CI | p-value |
| | Test vs. Untreated | x.xx | (x.xx, x.xx) | 0.xxxx |
| | Positive vs. Untreated | x.xx | (x.xx, x.xx) | 0.xxxx |

<sup>[1]</sup> From ANOVA on average rate over all raters including effects of treatment and age stratum.

<sup>[2]</sup> Difference is the first named treatment minus the second named treatment such that a positive difference favours the first named treatment

Page x of y



